CLINICAL TRIAL: NCT06606418
Title: Effect of Acupuncture for Rapid Eye Movement Sleep Behavior Disorder : a Randomized Controlled Trial
Brief Title: Effect of Acupuncture for Rapid Eye Movement Sleep Behavior Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wang Ziyi, Physician, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024BL02-085-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Rapid Eye Movement Sleep Behavior Disorder
Keywords: Rapid eye movement sleep behaviour disorder(RBD); acupuncture; randomized controlled trial; clinical research
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Active Comparator): The patients in this group received acupuncture treatment.
  Interventions: Other: Acupuncture group
- Sham acupuncture group (Sham Comparator): The patients in this group received sham acupuncture treatment.
  Interventions: Other: Sham acupuncture group

INTERVENTIONS:
Other: Acupuncture group — The patients in this group received acupuncture treatment 3 times a week for 4 weeks. Acupuncture points selection: bilateral Fei Shu (BL13), Xin Shu (BL15), Ji Shu (BL17), Gan Shu (BL18), PI Shu (BL20), Shen Shu (BL23), Shangqiu (SP5), Yin Bai (SP5), foot Qioyin (GB44), Li Dui (ST45). Acupuncture operation method: The patient took the lateral position and used Huacheng acupuncture needle (body length 40mm, diameter 0.30mm) to skew 0.5~0.8 inches at the back acupoint, 0.5~0.8 inches at Shangqiu (SP5), 0.1 inches at Yin Bai (SP5), foot Qiaoyin (GB44) and Li Dui (ST45), and left the needle for 30 minutes to wait for qi.
  Arms: Acupuncture group
Other: Sham acupuncture group — The patients in this group received sham acupuncture treatment 3 times a week for 4 weeks. Sham acupuncture points are selected at sham points close to the acupoints of the acupuncture group: 3 inches beside Fei Shu (BL13), Xin Shu (BL15), Ji Shu (BL17), Gan Shu (BL18), PI Shu (BL20), Shen Shu (BL23), 1 inches below Shangqiu (SP5), 0.1 inches behind the middle edge of the great toe, second toe and fourth toenail of the foot. Acupuncture operation method: The patient took the lateral position and used Huacheng acupuncture needle (body length 40mm, diameter 0.30mm) to pierce the skin shallowly, and left the needle for 30 minutes.
  Arms: Sham acupuncture group

SUMMARY:
Rapid eye movement (REM) sleep behaviour disorder (RBD) is a parasomnia that is characterized by abnormal behaviours occurring during REM sleep（a sleep stage）, often as dream enactments that can cause injury. Treatment options are limited. Pharmacological treatments include melatonin and clonazepam, but they have varying degrees of adverse reactions. Acupuncture is a green and safe means of treatment and has therapeutic value in sleep disorders. Using the theory of traditional Chinese medicine, the acupuncture treatment of RBD group points was formulated, and good clinical effect was obtained in the early clinical practice.This study was designed to explore the clinical efficacy of acupuncture in the treatment of RBD. Thirty patients with RBD who met the inclusion and exclusion criteria were randomly divided into acupuncture group and sham acupuncture group, and were subjected to a 2-week screening period, a 4-week treatment period, and a 2-week follow-up period.The investigators will primarily observe whether there is a reduction in the number of weekly RBD events recorded by the wCIRUS-RBD questionnaire before and after treatment, and the reduction in the RWA index recorded by video polysomnography (vPSG).

DETAILED DESCRIPTION:
Rapid eye movement (REM) sleep behaviour disorder (RBD) is a parasomnia that is characterized by abnormal behaviours occurring during REM sleep（a sleep stage）, often as dream enactments that can cause injury. Treatment options are limited. Pharmacological treatments include melatonin and clonazepam, but they have varying degrees of adverse reactions. Acupuncture is a green and safe means of treatment and has therapeutic value in sleep disorders. Using the theory of traditional Chinese medicine, the acupuncture treatment of RBD group points was formulated, and good clinical effect was obtained in the early clinical practice.This study was designed as a randomized, controlled and single-blind trial to explore the clinical efficacy of acupuncture in the treatment of RBD. Thirty patients with RBD who met the inclusion and exclusion criteria were randomly divided into acupuncture group and sham acupuncture group, and were subjected to a 2-week screening period, a 4-week treatment period, and a 2-week follow-up period.The investigators will primarily observe whether there is a reduction in the number of weekly RBD events recorded by the wCIRUS-RBD questionnaire before and after treatment, and the reduction in the RWA index recorded by video polysomnography (vPSG).

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients who meet the diagnostic criteria of ICSD-3. To confirm this diagnosis, one of the following conditions must be met: ① The diagnosis is RBD after previous vPSG examination. ② Those who have not been diagnosed should fill in RBDQ-HK. If the score is greater than 20, it indicates possible RBD, and accept vPSG test to confirm the diagnosis.
* (2)Patients belong to iRBD or secondary to the following three alpha-synuclein diseases: Parkinson's disease/multiple system atrophy/Lewy body dementia;
* (3) ≥18 years of age, male or female;
* (4) At least 2 episodes of RBD events in the past 2 weeks (recalled by the patient or described by family members), including: ① verbal behavior, such as Shouting and swearing; ② Physical movement behavior, such as waving arms, punching and kicking; ③Falling out of bed, dropping things around you, injuring yourself or others, which is speculated to be related to dreaming behavior;
* (5) Volunteer subjects and sign informed consent;
* (6) Can cooperate with the completion of this study.

Exclusion Criteria:

* (1) During pregnancy or lactation;
* (2) Patients with secondary RBD associated with narcolepsy or antidepressant use;
* (3) Patients with severe anxiety, depression and other mental diseases, alcohol abuse and/or psychoactive drug use, drug abusers and dependents;
* (4) Patients with serious underlying diseases, especially unstable diseases (such as malignant tumors, chronic obstructive pulmonary disease, unstable heart disease, etc.);
* (5) Patients with coagulation dysfunction, skin infection or damage at the surgical site should not receive acupuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
weekly CIRUS-RBD Questionnaire | Patients will be required to complete the wCIRUS-RBDQ questionnaire for a total of 8 weeks from the beginning of the screening period to the end of the follow-up period of 2 weeks after the end of treatment.
  The wCIRUS-RBDQ (weekly CIRUS-RBD Questionnaire) is used to record RBD-related information of patients every night of the week, and to be recalled and recorded by the patient and/or bed partner the next morning. Includes 4 items: (1) whether others know about your sleep; (2) Sleeping time; (3) whether there are vivid dreams, and if so, the frequency and severity of the dreams; (4) whether there is a dream deduction act, if so, what it is and how many times; The average weekly frequency of RBD events calculated in Part 4 of the questionnaire was used as the main outcome indicator. A higher frequency of RBD events means a worse outcome.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index(PSQI) | PSQI will be assessed before initiation of treatment and after 4 weeks of treatment.
  The Pittsburgh Sleep Quality Index (PSQI) is an international sleep assessment scale used to determine whether a person has sleep quality problems and their severity.The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. PSQI total score ≥7 points, can be judged as having sleep quality problems, PSQI score 7-11 points for mild, PSQI score 12-16 points for moderate, PSQI score 17-21 points for severe.
RBD Severity Scale (RBDss) | Assessment will be performed before initiation of treatment and after 4 weeks of treatment.
  The RBDss scale based on vPSG can be used to assess the RBD events and their severity, including motor events and vocal events. The results of RBDSS are divided into 8 points (0-3.5 points). Higher scores mean a worse outcome.
RWA index | Assessment will be performed before initiation of treatment and after 4 weeks of treatment
  REM sleep hypertonia (RWA) is the characteristic manifestation of BRD recorded by polysomngraphy (vPSG). The interpretation follows the AASM2.6 interpretation standard. The RWA index (The ratio of RWA frames to REM frames) can be detected by vPSG. Higher RWA index means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Huanqin Li, Physician, Principal Investigator — Beijing University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: The IPD used in the results publication will be avalible to researchers，in which the name of the patients and other Identity information will be hidden. They can access the IPD by contact the principal investigator through e-mail.